CLINICAL TRIAL: NCT00407628
Title: Neural Correlates of Lower Extremity Motor Recovery in Stroke Patients: Longitudinal Diffusion Spectrum Imaging Studies
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 9561703031; NSC95-2314-B-002-238-MY3
Record Dates: First submitted 2006-12-03; First posted 2006-12-05 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-01

CONDITIONS: Stroke
Keywords: Stroke; Diffusion spectrum tractography; Functional MRI (fMRI); Lower extremity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

SUMMARY:
To investigate the relationship between the integrity of the white matter, including the corticospinal tracts and the corpus callosum, with the recovery of lower extremity function in patients with cerebral stroke at the subacute and chronic stages.

DETAILED DESCRIPTION:
Recent studies have provided strong evidence that motor recovery after adult ischemic stroke is a function of neural plasticity. Up to date, it remains largely unknown as to the relationship between the integrity of the subcortical white matter with the lower extremity function recovery. Given the fact that the white matter is more resistant to ischemia after acute stroke than the gray matter (Falcao et al., 2004) and that the intensity of white matter in stroke has been found to be much greater in many brain areas in stroke than in healthy controls (Wen et al., 2004), it is of interest to study how the integrity of the subcortical white matter, primarily the corticospinal tracts and the corpus callosum, contributes to the recovery of lower extremity function in subacute and chronic stroke with lesions involving different areas of the brain.

ELIGIBILITY:
Inclusion Criteria:

* between 30 to 80 years old
* diagnosis of the first-time onset of stroke as confirmed by imaging studies
* within 30 days post onset University Hospital
* brain lesions mainly involving either the cortical primary motor cortex (M1) area or confined to the subcortical (M1 spared)
* No neurological or orthopedic problems which would affect their lower extremity function
* no contraindications for MRI studies

Exclusion Criteria:

* medically unstable
* unable to communicate with the experimenters

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: stroke patients
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2006-08; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
clinical assessments, included balance, motor, walking,ADL, will be obtained for tests performed on D7, D30 and D90 | D30, D90 and D180 post stroke onset

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Fang Tang, PhD, Study Chair — National Taiwan University Hospital
Locations (1):
- School and Graduate Institute of Physical Therapy College of Medicine, National Taiwan University, Taipei, Taiwan, China